CLINICAL TRIAL: NCT05070767
Title: Randomized Controlled Double Masked Two Arm Cross-over Study of Neurolenses in Subjects With Headaches
Brief Title: Neurolens Headache Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolens Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NLR - 210720
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Binocular Vision Disorder; Convergence Insufficiency; Headache; Computer Vision Syndrome
Keywords: headache; neurolenses; computer vision syndrome; convergence insufficiency; binocular vision; non-strabismic disorder; Digital vision syndrome
MeSH Terms: conditions — Ocular Motility Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Prospective randomized double masked two arm
Who Masked: Participant, Care Provider, Investigator
Masking Description: Prospective randomized double masked two arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Neurolens (Experimental): Our proprietary contoured prism lens design, commercially known as neurolens.
  Interventions: Device: Neurolens spectacle lens
- Control lens (Placebo Comparator): A simple refractive error correction lens
  Interventions: Device: Placebo spectacle lens

INTERVENTIONS:
Device: Neurolens spectacle lens — spectacle lens
  Arms: Neurolens
Device: Placebo spectacle lens — spectacle lens for refractive error correction
  Arms: Control lens

SUMMARY:
To understand the benefits of the neurolens Measurement Device and neurolens treatment as it pertains to treating symptoms related to Chronic Headaches. It is a Prospective randomized double masked two arm performed on a minimum of 200 to a maximum of 300 subjects identified as symptomatic (HIT-6 questionnaire score equal to or greater than 56) done across 3-15 clinical sites. There are two subgroups: a minimum of 100 in each subgroup (subgroup 1: pre-presbyopic (18-40 years); subgroup 2: presbyopic subjects (41-60 years).

DETAILED DESCRIPTION:
This study is a two-arm crossover study with two subgroups. Subjects will initially be assessed for their headache symptoms (Headache Impact Test (HIT-6) questionnaire) and then are provided an updated refractive prescription and will wear them for 35 ± 5 days. Symptoms will be reassessed after the 35-day control break in. If the subject's symptoms have subsided, they will be exited from the study and will keep their lenses. Provided the subject has symptoms (HIT questionnaire score ≥ 56) after their 35-day use of their updated prescription and they continue to meet the inclusion/exclusion criteria they will proceed to the evaluation portion of the protocol. The first arm receiving neurolens first and the second arm receiving the control first. The control is a single vision or PAL lens which yields the BCDVA and BCNVA of a test subject with no prismatic correction. The neurolens prescribed prism will be based on the practitioner's Rx using the subject's best response to a prism trial lens and must be within a half prism diopter of the neurolens value output of the neurolens Measurement Device and providing the subject's BCDVA and BCNVA. Participants will come back after 35 day wear of their first test lens and the symptom questionnaire is reassessed. They will be now be crossed over to the second pair of study lenses (i.e. subjects in the first arm will not receive control lens and the ones in the second arm will not receive neurolens). Participants will come back after 35 day wear of their second test lens and the symptom questionnaire is reassessed for the final time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, and between 18-60 years of age at the time of signing the informed consent.
* Best Corrected distance and near acuity are equal to or better than 20/25 Snellen Equivalent in each eye.
* Best Corrected distance and near binocular acuity are equal to or better than 20/25 Snellen Equivalent.
* Symptomatic as indicated by the HIT-6 questionnaire (Score equal to or greater than 56)
* Updated distance spectacle prescription must match the following

  a. Spherical power inclusive between +4.00D to -8.00D b. Cylinder power no more than -4.00Dcyl c. ADD power i. Subgroup 1: No ADD ii. Subgroup 2: minimum +1.00D ADD
* Subjects' eye alignment tests must match the following:

  a. Successful measurement on the neurolens Measurement Device (Acceptable MQI and a numerical neurolens Value, no Low MQI or Convergence Excess)
* Minimum stereo vision of 50 seconds of arc at 16 inches
* Capable of committing to the duration of the study.
* Willing to comply with study procedures

Exclusion Criteria:

* Subjects who need a vertical prism.
* Previously has worn neurolenses.
* Subjects who need a near add less than 1.00D
* Use of contact lenses during the study
* Lack of binocular vision, including strabismus, amblyopia, or suppression.
* Greater than 20 prism diopter of eye misalignment.
* Aniseikonia greater than 3.00D spherical equivalent difference between eyes
* Prior ocular surgery that in the estimation of the practitioner induces corneal scarring (RK, Corneal Transplant, etc.) or prior surgery involving the extraocular muscles (strabismus surgery). Surgeries that do not affect these parameters such as LASIK, PRK, or pterygium surgery are allowed.
* Anterior segment conditions that could obfuscate or obscure reflections from the cornea, or reduce visual acuity, including but not limited to corneal scarring, large pinguecula, pterygium, keratoconus, dermatochalasis, ptosis, exophthalmos or cataract.
* Clinical dry eye (defined as tear break-up time of less than 5 seconds)
* Intraocular pressures greater than 25 mmHg in either eye or uncontrolled glaucoma
* Macular disease, or any posterior segment finding which in the opinion of the investigator is visually and/or clinically significant
* Change in acute or prophylactic migraine treatment medication or dosage within the previous two months.
* Diabetes with ocular manifestation
* Previous head or neck trauma (for instance, car accident, etc.) requiring medical intervention.
* Open lesions or sores around the chin or eyes that will make contact with the device and may be subject to contraction or spread of infection.
* Physical tremors or muscle spasms that prevent a subject from sitting still.
* A history of seizures or seizure disorder.
* Women who are pregnant or lactating at the time of the study entry
* Mental incapacity that prevents a subject from being able to follow simple instructions such as "look at the target."

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test (HIT-6) questionnaire | 30-40 days
  Change in headache impact test (HIT-6) with the use of neurolenses compared to control lenses.
  The minimum response score for each question is 6 and the maximum is 13. Larger scores would indicate a more symptomatic patient.
  Larger difference in the cumulative response score between treatment visit and the baseline visit would indicate a greater impact of the treatment.

SECONDARY OUTCOMES:
Patients with reduced near point of convergence (NPC) | 30-40 days
  Change in the headache impact test (HIT-6) score with the use of neurolens compared to control lenses in subjects with reduced Near point of convergence (NPC).
  The minimum response score for each question is 6 and the maximum is 13. Larger scores would indicate a more symptomatic patient.
  Larger difference in the cumulative response score between treatment visit and the baseline visit would indicate a greater impact of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Van De Pol, OD PhD, Study Director — Neurolens Inc.
Locations (10):
- United States (10):
  - Advanced Vision and Achievement Center, Phoenix, Arizona
  - The Eye Center, Conyers, Georgia
  - Advanced Eyecare Center, Perry, Georgia
  - Eyecare of Rigby, Rigby, Idaho
  - Signature Eye Care, Lincoln, Nebraska
  - Buckeye Family Eye Clinic, Hillsboro, Ohio
  - Preferred Eye Care Center, Mt. Pleasant, South Carolina
  - Kapperman White and McGarvey, Chattanooga, Tennessee
  - Springhill Eye Care, Spring Hill, Tennessee
  - Eyes for Life, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will be providing a backend read-only excel spreadsheet of the raw data that was entered on the digital data platform provided to the clinical site.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available along with the publication for at least 5 years.
Access Criteria: On request